CLINICAL TRIAL: NCT02496637
Title: A Brief Appetite Awareness Intervention for Eating and Weight Regulation Among College Freshmen: A Randomized Clinical Trial
Brief Title: A Brief Appetite Awareness Intervention for Eating and Weight Regulation Among College Freshmen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1506S74643
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Eating Disorders
Keywords: Obesity; Eating Disorders; Appetite regulation; Eating Regulation
MeSH Terms: conditions — Obesity; Feeding and Eating Disorders | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Appetite Awareness (Experimental): Appetite Awareness Training (AAT) is an approach to increasing eating regulation through training individuals to eat in response to their appetite cues rather than external or emotional cues
  Interventions: Behavioral: Appetite Awareness
- Nutrition Education (Active Comparator): Nutrition education provides information about energy balance, dietary guidelines, portion and serving sizes, and other general dietary information.
  Interventions: Behavioral: Nutrition Education
- No Treatment Control (No Intervention): No intervention, assessment only

INTERVENTIONS:
Behavioral: Appetite Awareness — Appetite Awareness Training (AAT) is an approach to increasing eating regulation through training individuals to eat in response to their appetite cues rather than external or emotional cues
  Arms: Appetite Awareness
Behavioral: Nutrition Education — Nutrition education provides information about energy balance, dietary guidelines, portion and serving sizes, and other general dietary information.
  Arms: Nutrition Education

SUMMARY:
The proposed study is a randomized clinical trial investigating the effects of a weight gain and eating dysregulation prevention intervention among college freshmen women. It will compare Appetite Awareness Training (AAT) to a standard nutritional education group and a no treatment control group. Appetite Awareness Training approach to increasing eating regulation through training individuals to eat in response to their appetite cues rather than external or emotional cues.

DETAILED DESCRIPTION:
All female freshmen students residing in the university dorms were recruited to participate in this study. After completing the baseline assessment, eligible participants were randomly assigned to one of the three arms. Those in the AAT condition received guided administration of AAT over the course of three weekly group sessions, with an additional booster session three weeks after completion (week 6). The standard treatment comparison group received four similarly timed group sessions of psychoeducational/nutrition information facilitated by a registered dietician. A manualized approach to administration of the intervention was created based on the AAT treatment and was strictly followed in order to standardize the implementation of the prevention groups. The no-treatment control group only participated in the assessments.

ELIGIBILITY:
Inclusion Criteria:

* Incoming University of Minnesota Duluth freshmen women residing in on campus dormitories

Exclusion Criteria:

* Males, non-dormitory residing, non-freshmen.

Ages: 18 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight measured in pounds | Baseline, 6 weeks, 4 months
Change in Appetite Awareness as assessed by the Interoceptive Awareness Questionnaire (appetite subscale) | Baseline, 6 weeks, 4 months

SECONDARY OUTCOMES:
Change in Body Image as assessed by the Satisfaction and Dissatisfaction with Body Parts Scale | 6 weeks, 4 months
Change in Weight Management self-efficacy as assessed by the Weight Efficacy Lifestyle Questionnaire | 6 weeks, 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Lara LaCaille, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Duluth, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No